CLINICAL TRIAL: NCT03673995
Title: Use of Myoinositol Plus L-tyrosine, Selenium and Chromium in PCOS Women
Brief Title: Myoinositol Plus L-tyrosine, Selenium and Chromium in PCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pharmarte srl (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PharmarteLtyrosine1
Record Dates: First submitted 2018-08-22; First posted 2018-09-17 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2018-09

CONDITIONS: Polycystic Ovary Syndrome; Menstrual Problem; Hirsutism
MeSH Terms: conditions — Polycystic Ovary Syndrome; Menstruation Disturbances; Hirsutism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Myo-inositol+L-tyrosine (Experimental): One sachet per day containing 2000 mg myo-inositol, 500 mg L-tyrosine, 40 mcg chromium picolinate, 55 mcg selenium, 200 mcg folic acid for improving PCOS symptoms.
  Interventions: Dietary Supplement: Myo-inositol+L-tyrosine

INTERVENTIONS:
Dietary Supplement: Myo-inositol+L-tyrosine — PCOS patients were treated every day, with one sachet containing 2000 mg myo-inositol, 500 mg L-tyrosine, 40 mcg chromium picolinate, 55 mcg selenium, 200 mcg folic acid. All patients underwent, before starting the therapy, after 3 months and 6 months, hormonal, hirsutism and ovulation assesment.

SUMMARY:
PCOS patients were treated every day, with one sachet containing 2000 mg myo-inositol, 500 mg L-tyrosine, 40 mcg chromium picolinate, 55 mcg selenium, 200 mcg folic acid. All patients underwent, before starting the therapy, after 3 months and 6 months, hormonal evaluation , hirsutism scoring and ovulation assesment. Most of them during the treatment improved their symptoms.

ELIGIBILITY:
Inclusion Criteria:

° PCOS patients

Exclusion Criteria:

* thyroid dysfunction
* hyperprolactinemia
* adrenal hyperplasia
* patients taking oral contraceptive
* any other endocrinological pathologies

Ages: 16 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 186 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2018-08-22 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Restore of regular menstrual period | 6 months of treatment
  Self report

SECONDARY OUTCOMES:
Improving hirsutism | 6 months of treatment
  Standardised visual scales are preferred when assessing hirsutism, such as the modified Ferriman Gallwey score (mFG) with a level ≥ 4 - 6 indicating hirsutism,
Restore ovulation | 6 months of treatment
  Progesterone value in luteal phase

CONTACTS AND LOCATIONS:
Overall Officials: Mario Montanino Oliva, M.D., Principal Investigator — Altamedica Reproductive Medicine
Locations (1):
- Altamedica Reproductive Medicine, Roma, Italy